CLINICAL TRIAL: NCT03734965
Title: The Comparison of Awake Fiberoptic And Awake Video Laryngoscopy Tracheal
Brief Title: The Comparison of Awake Fiberoptic And Awake Video Laryngoscopy Tracheal Intubation in Cervical Surgery
Acronym: TCAFAVLTICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Fatih Sag, Principal Investigator; Resident Doctor, Trakya University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TÜTF-BAEK 2018/90
Record Dates: First submitted 2018-10-19; First posted 2018-11-08 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Cervical Disorder
Keywords: aweken intubation; fiberoptic; videolaryngoscopy
MeSH Terms: conditions — Uterine Cervical Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWAKEN INTUBATION FIBEROPTIC (Active Comparator): awaken intubation
  Interventions: Device: AWAKEN INTUBATION
- AWAKEN INTUBATION VIDEOLARYNGOSCOPY (Experimental): awaken intubation
  Interventions: Device: AWAKEN INTUBATION

INTERVENTIONS:
Device: AWAKEN INTUBATION — Intubation

SUMMARY:
Intubation processes of patients under general anesthesia are important in terms of patient morbidity and mortality. The cervical region has also anatomical and physiologic speciality in which stability of the general condition of the patient during this intubation process. The cervical region needs to be manipulated very carefully due to respiratory center, cardiovascular balance and neurological integrity. During general anesthesia, the patient will be under the effect of muscle relaxant and especially the cervical region becomes vulnerable to trauma. The intubations made by affecting the cervical region as little as possible change the morbidity and mortality. Intubation with fiberoptic bronchoscopy and videolaryngoscopy has reduced the complications that other methods can cause. Awake intubation with fiberoptic bronchoscopy and videolaryngoscopy is important for neurological evaluation during the procedure. In this study, we aimed to compare awake intubation by videolaringoscopy and fiberotic bronchoscopy in patients with intubation difficulties due to restriction of neck movements in cervical surgery.

DETAILED DESCRIPTION:
INTRODUCTION: Intubation processes of patients under general anesthesia are important in terms of patient morbidity and mortality. The cervical region has also anatomical and physiologic speciality in which stability of the general condition of the patient during this intubation process. The cervical region needs to be manipulated very carefully due to respiratory center, cardiovascular balance and neurological integrity. During general anesthesia, the patient will be under the effect of muscle relaxant and especially the cervical region becomes vulnerable to trauma. The intubations made by affecting the cervical region as little as possible change the morbidity and mortality. Intubation with fiberoptic bronchoscopy and videolaryngoscopy has reduced the complications that other methods can cause. Awake intubation with fiberoptic bronchoscopy and videolaryngoscopy is important for neurological evaluation during the procedure. In this study, we aimed to compare awake intubation by videolaringoscopy and fiberotic bronchoscopy in patients with intubation difficulties due to restriction of neck movements in cervical surgery.

METHODS: Patients in the ASA I-II-III risk group, aged 18-80 years, who will undergo cervical surgery operation between 01.04.2018 and 01.04.2020 by the Brain and Neurosurgeon at Trakya University Medical Faculty Hospital will be included. Patients will be prospectively randomized into 2 groups; Group F (intubation with fiberoptic in awake patients), Group V (intubation with videolaringoscopy in awake patients). In successful intubations the time between the time of access to the criterion laryngoscope and the appearance of the vocal cord will be assumed to be 60 seconds. Complications during intubation (mucosal injury, tooth trauma, lip injury, hypoxia (SpO2 <95%) and esophageal intubation) will be recorded. After intubation, the presence of blood in the Endotracheal Tube (ETT) or sore throat, which is expressed by the patient after recovery, will also be recorded.

STATISTICAL METHODS: Student-T test or Mann Whitney U test will be applied among the groups. Ki-Kara test will be used to compare categorical data.

CONCLUSION: Evaluation of mortality and morbidity of the patients awake intubation with fiberoptic bronchoscopy and videolaryngoscopy for cervical trauma surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years who planning cervical surgery

Exclusion Criteria:

* Patients with motor and sensory loss,
* Congenital neurological deficits, those with fiberoptic intubation inconveniences (with cerebrovascular case and hypertension),
* Patients with awake intubation (neuropsychiatric patients with orientation and cooperativeness impairment),
* Cardiovascular patients with local anesthetic allergy,
* Patients with difficult intubation history,
* Cervical surgery,
* Body mass index> 30 kg / m2,
* Mallampati score III-IV,
* Thyromental distance> 6 cm,
* Risk of gastric aspiration and pregnancies will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
awaken intubation | It is 60 seconds for succesfully intubation on procedure from it is starting to completed tracheal intubation
  succesful intubation

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap Hekimoglu Sahin, Proffesor, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No